CLINICAL TRIAL: NCT07081841
Title: Long-Term Safety and Efficacy Follow-up of AB-1005 Gene Transfer Study Participants With Parkinson's Disease or Multiple System Atrophy
Brief Title: AB-1005 Long-Term Follow-up Study
Status: Enrolling by invitation | Type: Observational
Sponsor: AskBio Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: ASK-PD0-CS002
Record Dates: First submitted 2025-06-09; First posted 2025-07-23 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Parkinson's Disease; Multiple System Atrophy, Parkinson Variant
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with PD
  Interventions: Other: Observation
- Participants with MSA-P
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — This is an observational study in which safety laboratories and non-invasive routine clinical assessments are conducted to gauge long term safety and efficacy.

SUMMARY:
This is an observational, long term, follow-up study for participants with Parkinson's disease (PD) or Multiple System Atrophy-Parkinsonian subtype (MSA-P) who participated in prior interventional studies with AB-1005. It is intended to better understand the long-term safety of AB-1005, how well tolerated it is and how long lasting the effects are.

ELIGIBILITY:
Inclusion Criteria:

* PD and MSA-P participants that are or were enrolled in an interventional AB-1005 study and provide informed consent

Exclusion Criteria:

* There are no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who have participated in interventional studies of AB-1005.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2037-09-30 (Estimated); Study Completion 2038-03-30 (Estimated)

PRIMARY OUTCOMES:
Long term safety and tolerability | Up to 10 years post surgery
  Measure of the occurrence of serious and non-serious adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No